CLINICAL TRIAL: NCT02635685
Title: Clinical Decision Support for Stroke Prevention in Atrial Fibrillation - a Cluster Randomized Trial in the Primary Care Setting
Brief Title: Clinical Decision Support for Stroke Prevention in Atrial Fibrillation
Acronym: CDS-AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Linkoeping (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Lars Karlsson, MD, PhD, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015/398-32
Record Dates: First submitted 2015-11-18; First posted 2015-12-21 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Cardiovascular Disease; Atrial Fibrillation; Stroke
Keywords: Atrial fibrillation; Stroke; Clinical Decision Support; Anticoagulants
MeSH Terms: conditions — Cardiovascular Diseases; Atrial Fibrillation; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Intervention with Clinical Decision Support tool installed on units.
  Interventions: Other: Clinical Decision Support tool
- Control group (No Intervention): Control group without intervention with Clinical Decision Support tool installed on units.

INTERVENTIONS:
Other: Clinical Decision Support tool — Automatized support tool for identification of patients with a diagnosis of atrial fibrillation without appropriate anticoagulant therapy for stroke prevention.
  Arms: Intervention group

SUMMARY:
A cluster randomised study in the primary care setting to evaluate a electronic clinical decision tool for stroke prophylaxis in patients with atrial fibrillation.

DETAILED DESCRIPTION:
Atrial fibrillation is the most common form of arrhythmia, affecting more than three percent of the population. The condition carries an increased risk of thromboembolism, in particular stroke. In 2013 approximately 25000 acute strokes were diagnosed in Sweden, with the result of death or severe disability in nearly half of the cases. Numerous studies have shown that the risk for stroke can be reduced by approximately 60-70 % with the use of anticoagulant therapy to patients with one or several risk factors for stroke and concurrent atrial fibrillation. The European Society of Cardiology recommends use of the CHA2DS2VASc algorithm to identify persons at increased risk for stroke in the setting of atrial fibrillation. Prophylaxis is recommended if CHA2DS2VASc ≥ 1 (not only female gender).

The agents used include warfarin and the more recently developed non-vitamin k oral anticoagulants (NOACs). Despite good evidence and recommendations in current guidelines, however, there remains a substantial undertreatment in this group of patients.

The Swedish Association of Local Authorities and Regions have shown that only 63% of patients with a CHA2DS2VASc score ≥ 2 are prescribed anticoagulant therapy [7]. The reasons for this is most likely multifactorial, including ignorance of the CHA2DS2VASc algorithm as well as reluctance of the use of potent drugs from both doctors and patients. Furthermore, the high pace in modern medicine increase the risk of missing the diagnosis of atrial fibrillation and/or the conditions constituting the CHA2DS2VASc algorithm.

Clinical decision tools is a relatively new phenomena in modern medicine showing promising results, but evidence for clinical outcome are sparse. The clinical decision tool for stroke prevention (CDSS) has been developed in collaboration between Cambio Cosmic (the supplier of the electronic journal in the county of Östergötland), the Cardiology Department at Linköping University hospital and primary care professionals. The decision tool is activated when a patient is being logged into the electronic journal. If the patient has a diagnosis of atrial fibrillation (or atrial flutter) and a CHA2DS2VASc score ≥ 1 (not only female gender) without current anticoagulant therapy, a screen warning will appear. By clicking on the warning, the responsible physician will get an overview of the patient's diagnosis according to the CHA2DS2VASc algorithm. Furthermore, a calculation of the estimated stroke risk for the coming year will appear, and links to national guidelines be provided. The physician can thereafter decide to prescribe anticoagulant therapy in accordance with current guidelines or, alternatively, postpone the decision/make a decision to refrain from medication. In case the choice is made to refrain from medication the physician is asked to choose between a set of predetermined reasons in order to monitor the main reasons for deviation from guidelines.

If, on the other hand, the patient has anticoagulant therapy in accordance with current guidelines, no screen warning will appear.

CDSS has shown promising results in a pilot study conducted at five units in the County of Östergötland during the fall of 2014. The aim of the present study is to investigate this computerized decision tool in a large randomized trial in the primary care setting.

Study design The present study is a cluster randomized study in the primary care setting in the County of Östergötland, Sweden. The investigators intend to include all primary care units (n = 43) in the County of Östergötland. Participation is non-compulsory. The population in the County of Östergötland is 442 105 (December 2014)

At the time of inclusion all primary care units will be stratified in four strata based on the number of patients listed on each unit and current adherence to guidelines (i.e. the percentage of patients with a diagnosis of atrial fibrillation and CHA2DS2VASc ≥ 1 (not only female gender) that are currently prescribed anticoagulant therapy). They will thereafter be randomized to intervention with the CDSS application or serve as a control unit (continue with usual care, randomized 1:1). Prior to randomization all the participating general practitioners will receive an education about atrial fibrillation and the associated risk of stroke, including the CHA2DS2VASc algorithm and an overview of anticoagulant therapy. Furthermore, all units receiving the CDSS will have a briefing about the technical aspects of using the application.

ELIGIBILITY:
Inclusion Criteria:

* Primary care centers in the county of Östergötland, Sweden.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 442105 (Actual)
Dates: Start 2016-01-11 (Actual); Primary Completion 2017-01-11 (Actual); Study Completion 2025-01-11 (Estimated)

PRIMARY OUTCOMES:
Adherence to guidelines defined as the percentage of patients with atrial fibrillation and CHA2DS2VASc ≥ 1, (not only female gender) that are prescribed anticoagulant therapy (ATC-code B01A). | 12 months after study commencement
  The data will be recorded through the electronic journal where the diagnosis for atrial fibrillation/flutter, the conditions constituting the CHA2DS2VASc algorithm as well as the medication list is logged.

SECONDARY OUTCOMES:
Reduction av thromboembolism. This will be analyzed through the electronic medical journal by identifying the patients with new (since commencement of the study) diagnosis of thromboembolism. ICD-10 codes I63-64, G45, I75 will be analyzed. | 12 months after study commencement and 3 and 6 years after study finish.
Analysis of physician acceptance of a clinical decision tool in the primary care setting with questionnaires to randomly assigned general physicians. | Before study commencement and after 12 months
  The extended Technology Acceptance Model is implemented with modifications in order to capture moderating factors of acceptance.
Analysis of reasons to deviate from guidelines. As part of the clinical decision tool there are prespecified reasons to choose from if no therapy is prescribed. The main reasons will be summarized. | 12 months after study commencement
Cost-effectiveness of using clinical decision support tool for stroke prevention in the primary care setting. | 12 months follow-up
  : Resource use regarding education of general practitioners and the time for using the clinical decision support tool is going to be identified and translated into healthcare costs by assigning a unit cost.
  Cost of the clinical decision support tool is also included to get the mean healthcare cost/patient.
  The effectiveness measure is percentage of all patients with atrial fibrillation getting anticoagulation therapy in the clinical decision support tool group compared with the control group.
  This is a trial based evaluation. We will also calculate longterm results with a modelling approach.

CONTACTS AND LOCATIONS:
Overall Officials: Lars O Karlsson, MD, PhD, Principal Investigator — Department of Cardiology and Department of Medical and Health Sciences, Linköping University, Linköping, Sweden
Locations (1):
- The County of Östergötland, Linköping, Sweden

REFERENCES:
- [Background] Friberg L, Bergfeldt L. Atrial fibrillation prevalence revisited. J Intern Med. 2013 Nov;274(5):461-8. doi: 10.1111/joim.12114. Epub 2013 Aug 7. PMID 23879838
- [Background] Riks-stroke. Annual report 2013 (in Swedish). http://www.riksstroke.org/wp-content/uploads/2014/07/Strokerapport_AKUTTIA3man_LR.pdf. Accessed November 2014.
- [Background] Hart RG, Pearce LA, Aguilar MI. Meta-analysis: antithrombotic therapy to prevent stroke in patients who have nonvalvular atrial fibrillation. Ann Intern Med. 2007 Jun 19;146(12):857-67. doi: 10.7326/0003-4819-146-12-200706190-00007. PMID 17577005
- [Background] Camm AJ, Lip GY, De Caterina R, Savelieva I, Atar D, Hohnloser SH, Hindricks G, Kirchhof P; ESC Committee for Practice Guidelines-CPG; Document Reviewers. 2012 focused update of the ESC Guidelines for the management of atrial fibrillation: an update of the 2010 ESC Guidelines for the management of atrial fibrillation--developed with the special contribution of the European Heart Rhythm Association. Europace. 2012 Oct;14(10):1385-413. doi: 10.1093/europace/eus305. Epub 2012 Aug 24. No abstract available. PMID 22923145
- [Background] Bjorck S, Palaszewski B, Friberg L, Bergfeldt L. Atrial fibrillation, stroke risk, and warfarin therapy revisited: a population-based study. Stroke. 2013 Nov;44(11):3103-8. doi: 10.1161/STROKEAHA.113.002329. Epub 2013 Aug 27. PMID 23982711
- [Background] Kakkar AK, Mueller I, Bassand JP, Fitzmaurice DA, Goldhaber SZ, Goto S, Haas S, Hacke W, Lip GY, Mantovani LG, Turpie AG, van Eickels M, Misselwitz F, Rushton-Smith S, Kayani G, Wilkinson P, Verheugt FW; GARFIELD Registry Investigators. Risk profiles and antithrombotic treatment of patients newly diagnosed with atrial fibrillation at risk of stroke: perspectives from the international, observational, prospective GARFIELD registry. PLoS One. 2013 May 21;8(5):e63479. doi: 10.1371/journal.pone.0063479. Print 2013. PMID 23704912
- [Background] Öppna jämförelser: hälso- och sjukvård 2014, del 2 (in Swedish). http://webbutik.skl.se/sv/artiklar/oppna-jamforelser-halso-och-sjukvard-2014-del-1.html. Accessed December 4, 2014.
- [Background] Lobach D, Sanders GD, Bright TJ, Wong A, Dhurjati R, Bristow E, Bastian L, Coeytaux R, Samsa G, Hasselblad V, Williams JW, Wing L, Musty M, Kendrick AS. Enabling health care decisionmaking through clinical decision support and knowledge management. Evid Rep Technol Assess (Full Rep). 2012 Apr;(203):1-784. PMID 23126650
- [Background] Bright TJ, Wong A, Dhurjati R, Bristow E, Bastian L, Coeytaux RR, Samsa G, Hasselblad V, Williams JW, Musty MD, Wing L, Kendrick AS, Sanders GD, Lobach D. Effect of clinical decision-support systems: a systematic review. Ann Intern Med. 2012 Jul 3;157(1):29-43. doi: 10.7326/0003-4819-157-1-201207030-00450. PMID 22751758
- [Derived] Persson Lindell O, Henriksson M, Karlsson LO, Nilsson S, Charitakis E, Janzon M. Cost-effectiveness of a clinical decision support system for atrial fibrillation: an RCT-based modelling study. Eur Heart J Digit Health. 2025 Aug 1;6(5):997-1005. doi: 10.1093/ehjdh/ztaf087. eCollection 2025 Sep. PMID 40984984
- [Derived] Karlsson LO, Nilsson S, Bang M, Nilsson L, Charitakis E, Janzon M. A clinical decision support tool for improving adherence to guidelines on anticoagulant therapy in patients with atrial fibrillation at risk of stroke: A cluster-randomized trial in a Swedish primary care setting (the CDS-AF study). PLoS Med. 2018 Mar 13;15(3):e1002528. doi: 10.1371/journal.pmed.1002528. eCollection 2018 Mar. PMID 29534063